CLINICAL TRIAL: NCT06264830
Title: Comparing the Effect of Depth of Focus Difference in High Myopic Patients Receiving Cataract Operations Between 3D Visualization System and Traditional Optical Microscope.
Brief Title: 3D Visualization System in Highly Myopic Cataract Operation
Acronym: 3D-HiMCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202307103DIPC
Record Dates: First submitted 2024-01-21; First posted 2024-02-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Cataract; High Myopia
Keywords: Cataract; High Myopia; Digital 3D System; Depth of Field
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional-binocular-microscope-assisted standard cataract operation (Active Comparator): In this group, patients undergo standard modern cataract operation during which the surgeon use conventional binocular microscope
  Interventions: Procedure: Standard cataract operation
- Alcon-NGENUITY® (NG)-System-assisted standard cataract operation (Experimental): In this group, patients undergo standard modern cataract operation during which the surgeon use the Alcon NGENUITY® (NG) System
  Interventions: Device: Alcon-NGENUITY®(NG)-system; Procedure: Standard cataract operation

INTERVENTIONS:
Device: Alcon-NGENUITY®(NG)-system — During operation, the Alcon NGENUITY® (NG) System is mounted on microscope, while the surgeon will wear 3D glasses, watch 3D screen, and perform operation
  Arms: Alcon-NGENUITY® (NG)-System-assisted standard cataract operation
Procedure: Standard cataract operation — Standard, modern cataract extraction with standard phacoemulsification technique, and posterior chamber intraocular lens implantation.

SUMMARY:
This study aims to investigate the impact of depth of field differences between the use of the 3D imaging system (NGENUITY® 3D Visualization System, Alcon, TX, USA) and conventional optical microscope in cataract surgery for highly myopic patients on intraoperative parameters and outcomes.

DETAILED DESCRIPTION:
The objective of this study is to compare the surgical outcomes and parameters between cataract surgeries performed using the NGENUITY® 3D Visualization System (Alcon, TX, USA), a 3D imaging system, and the current standard binocular microscope in highly myopic patients. The focus is on evaluating the differences in depth of field and their impact on intraoperative parameters and outcomes.

This prospective randomized controlled trial aims to enroll patients with both high myopia and cataracts requiring surgical intervention. Participants will be randomly assigned to undergo cataract surgery using the current standard binocular microscope (control group) or the NGENUITY® 3D Visualization System (Alcon, TX, USA) (study group). The study will compare intraoperative parameters, surgical outcomes, and the incidence of potential complications, including the frequency of microscope adjustments during surgery, total distance of adjustments during surgery, distance needed to achieve clear focus from the corneal surface to the posterior capsule, surgical duration, cumulative ultrasound energy during surgery, and occurrence of surgical complications.

ELIGIBILITY:
Inclusion Criteria:

1. High myopia (axial length of 26 millimeters or more).
2. Presence of clinically significant age-related nuclear cataract requiring surgery, assessed using the International Classification System for Cataract (Lens Opacities Classification System III, LOC III), with a graded score indicating nuclear cataract (LOC III NC/NO grade 3-5).
3. Participants must be 20 years of age or older.

Exclusion Criteria:

1. The target eye has undergone vitrectomy surgery.
2. The target eye has undergone corneal refractive surgery.
3. Presence of corneal diseases such as corneal dystrophy, corneal trauma, corneal scarring, corneal ulcers, or clinically significant corneal softening that significantly affects the clarity of cataract surgery.
4. Complicated cataracts with features such as extreme hardness, complex composition, zonular laxity, lens dislocation, extensive capsular fibrosis, or those falling under the international cataract classification standards LOCIII NO/NC6 or C4-C5 or P4-P5.
5. Presence of other non-myopia-related eye diseases significantly affecting the complexity of surgery, such as adhesive uveitis causing adhesions, corneal damage due to trauma or lens dislocation, structural changes and adhesions due to intraocular inflammation, or severe uncorrected strabismus affecting eye alignment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of times of Microscopic focus adjustment, measured by counting from the video recordings | Throughout operation
  A video recorder will focus on the sliding joint between main suspension arm of microscope and its lens system. Once the surgeon change the focus, the marks on both side of the joint will change their relative positions. The times of changes will be counted from the video recording.
Total moving distance in millimeter of microscope-lens-system relative to suspension arm, measured by ruler set on microscope | Throughout operation
  On the microscope one ruler will place on the suspension arm of microscope just beside the sliding joint of main optic lens system. On the side of main optic lens system, there will be a mark. When the surgeon change the focus of microscope. The mark will change its position relative to the ruler with millimeter in scale. The total moving distance is the add-ups of all changes during operation in absolute value.
Distance of subjective focus change in millimeter between corneal surface and surface of posterior capsule, measured by ruler set on microscope | During the operation, immediately after lens material is removed, and immediately before the intraocular lens is implanted.
  On the microscope one ruler will place on the suspension arm of microscope just beside the sliding joint of main optic lens system. On the side of main optic lens system, there will be a mark. When the surgeon change the focus of the microscope. The mark will change its position relative to the ruler with millimeter in scale. Distance in millimeter of subjective focus between corneal surface and surface of posterior capsule can thus be measured.

SECONDARY OUTCOMES:
Total operation time | Throughout operation
  Total operation time
Cumulative dissipated energy (CDE) of phacoemulsification, that is automatically measured and demonstrated on the screen of phacoemulsification machine (Centurion) | Throughout operation
  Cumulative dissipated energy (CDE) is defined as mean phaco power times phaco time. CDE will be automatically measured and calculated by the Alcon centurion phacoemulsification machine, and will be demonstrated on the screen of the machine. CDE is itself the unit. The lower the CDE for an operation, the better.
Number of Participants with intraoperative complication | Throughout operation
  Number of Participants with intraoperative complication
Best-corrected visual acuity of the operated eye of Participants at each postoperative follow-up within 3 month, measured with Snellen chart under standard condition (6 meters in distance and standard illumination of environment) | Within 3 month after operation, at postoperative day1, at postoperative week 1, at post operative month 1, at post operative month 3
  The best-corrected visual acuity (BCVA) measured with Snellen chart is expected to range from 20/20(1.0) to 20/400(0.05). The refraction of the eye will be carefully corrected using trial lens. The higher the Snellen-chart value, and better the vision. For worse vison. The BCVA will be documented with able to count finger at certain distance ( such as100 centimeter or 30 centimeter). For even worse one, the BCVA will be documented with able to tell hand waving or not at certain distance ( such as100 centimeter or 30 centimeter). For even worse one, the BCVA will be documented with light perception or no light perception.
Number of Participants with post-operative complication | Within three month after operation, at postoperative day1, at postoperative week 1, at post operative month 1, at post operative month 3
  Number of Participants with post-operative complication
Intraocular pressure of the operated eye of participants at each postoperative follow-up within 3 month, measured with pneumatic tonometer | Within 3 month after operation, at postoperative day1, at postoperative week 1, at post operative month 1, at post operative month 3
  The intraocular pressure will be measured with pneumatic tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Tzyy-Chang Ho, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamasaki I, Shibata K, Shimizu T, Kono R, Morizane Y, Shiraga F. Lights-out Surgery for Strabismus Using a Heads-Up 3D Vision System. Acta Med Okayama. 2019 Jun;73(3):229-233. doi: 10.18926/AMO/56865. PMID 31235970
- [Background] Weinstock RJ, Diakonis VF, Schwartz AJ, Weinstock AJ. Heads-up Cataract Surgery: Complication Rates, Surgical Duration, and Comparison With Traditional Microscopes. J Refract Surg. 2019 May 1;35(5):318-322. doi: 10.3928/1081597X-20190410-02. PMID 31059581
- [Background] Kita M, Mori Y, Hama S. Hybrid wide-angle viewing-endoscopic vitrectomy using a 3D visualization system. Clin Ophthalmol. 2018 Feb 12;12:313-317. doi: 10.2147/OPTH.S156497. eCollection 2018. PMID 29491704
- [Background] Skinner CC, Riemann CD. "HEADS UP" DIGITALLY ASSISTED SURGICAL VIEWING FOR RETINAL DETACHMENT REPAIR IN A PATIENT WITH SEVERE KYPHOSIS. Retin Cases Brief Rep. 2018 Summer;12(3):257-259. doi: 10.1097/ICB.0000000000000486. PMID 27841831
- [Background] Coppola M, La Spina C, Rabiolo A, Querques G, Bandello F. Heads-up 3D vision system for retinal detachment surgery. Int J Retina Vitreous. 2017 Nov 20;3:46. doi: 10.1186/s40942-017-0099-2. eCollection 2017. PMID 29188074
- [Background] Wai YZ, Fiona Chew LM, Mohamad AS, Ang CL, Chong YY, Adnan TH, Goh PP. The Malaysian cataract surgery registry: incidence and risk factors of postoperative infectious endophthalmitis over a 7-year period. Int J Ophthalmol. 2018 Oct 18;11(10):1685-1690. doi: 10.18240/ijo.2018.10.17. eCollection 2018. PMID 30364221
- [Background] Qian Z, Wang H, Fan H, Lin D, Li W. Three-dimensional digital visualization of phacoemulsification and intraocular lens implantation. Indian J Ophthalmol. 2019 Mar;67(3):341-343. doi: 10.4103/ijo.IJO_1012_18. PMID 30777950
- [Background] Ramirez Mejia M, Arroyo Munoz L, Medina Perez AB, Mendoza Velasquez C, Ceja Martinez J, Camacho Ordonez A, Guerrero-Berger O. Magnification and Refocusing Comparison in Cataract Surgery Using a Heads-Up Three-Dimensional Visualization System versus Conventional Binocular Microscopy. Clin Ophthalmol. 2023 Aug 15;17:2333-2339. doi: 10.2147/OPTH.S423372. eCollection 2023. PMID 37600146
- [Background] Kelkar JA, Kelkar AS, Bolisetty M. Initial experience with three-dimensional heads-up display system for cataract surgery - A comparative study. Indian J Ophthalmol. 2021 Sep;69(9):2304-2309. doi: 10.4103/ijo.IJO_231_21. PMID 34427206
- [Background] Liu J, Wu D, Ren X, Li X. Clinical experience of using the NGENUITY three-dimensional surgery system in ophthalmic surgical procedures. Acta Ophthalmol. 2021 Feb;99(1):e101-e108. doi: 10.1111/aos.14518. Epub 2020 Jul 9. PMID 32643263